CLINICAL TRIAL: NCT06653569
Title: A Swiss Multi-center, Randomized, Placebo-controlled Trial on the Efficacy of Baloxavir Marboxil to Reduce Time to Clinical Improvement in Adult Patients Hospitalized for Influenza
Brief Title: Efficacy of Baloxavir Against Influenza in Hospitalized Patients: the INFLUENT Study (INpatients InFLUENza Treatment)
Acronym: INFLUENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dre Pauline Vetter (Other)
Collaborators: Swiss National Science Foundation (Other); University Hospital, Geneva (Other); University of Geneva, Switzerland (Other); Ente Ospedaliero Cantonale, Ticino, Switzerland (Other); Centre Hospitalier Universitaire Vaudois (Switzerland) (Unknown); Universitätspital Zürich, (Switzerland) (Unknown); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Dre Pauline Vetter, Senior staff physician, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-01535; 33IC30_221790 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Influenza Disease; Flu
Keywords: antiviral treatment; baloxavir marboxil; influenza complications; hospitalization; severe influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Intervention Model Description: Placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- antiviral treatment (Experimental): baloxavir marboxil
  Interventions: Drug: Baloxavir Marboxil
- placebo (Placebo Comparator): Pacebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baloxavir Marboxil — The antiviral baloxavir marboxil administered in one unique dose.
  1 capsule (40 mg) if participant weighs < 80 kg; 2 capsules (80 mg) if participant weighs ≥ 80 kg
  Arms: antiviral treatment
Drug: Placebo — Patients in the placebo group will receive one unique dose of placebo. 1 capsule if participant weighs < 80 kg; 2 capsules (80 mg) if participant weighs ≥ 80 kg.
  Arms: placebo

SUMMARY:
The purpose of this clinical trial is to find out if the medication called baloxavir marboxil (sold under the brand name Xofluza®) can help to reduce the time needed to recover from flu when patients need an hospitalization. Patients infected by influenza and requiring a hospitalization will be approched to be included in the study.

The main questions are:

1. When someone is hospitalized with a severe influenza infection, does baloxavir help to reduce the time needed to recover?
2. Can baloxavir marboxil help to shorten the amount of time people need to stay in the hospital with severe flu?
3. Can baloxavir marboxil help to reduce the risk of life-threatening complications as well as of death due to severe flu?
4. Can baloxavir reduce duration of contagiousness?

To be able to measure the above, the investigators will compare two groups of patients: One group receiving baloxavir marboxil, the other group receiving a mock treatment called placebo.

Participants will:

* Take one single dose of baloxavir marboxil or placebo soon after hospitalization.
* Vital signs will be followed three times per day during hospital stay.
* Have a nose swab to detect the presence of influenza virus on the first and third day of trial participation.
* Answer to a short quality of life questionnaire on the phone 3 months after receiving the study treatment.

DETAILED DESCRIPTION:
Background: Influenza virus is a major source of seasonal outbreaks and is the leading candidate for a future pandemic. Each winter thousands of people are hospitalized with infection complications. The most at risk are the very young (< 5 years), the elderly (>65 years old) and those with a weak immune system. When a person is hospitalized because of the flu, it is not always clear if the administration of a specific medicine that fights the virus (called an antiviral) will help.

Most studies looked at antivral drug benefits among people with mild flu, who didn't need to be hospitalized. They found that if the antiviral is started early (up to two days after the symptoms started), it can make the symptoms go away a little faster. But for people in the hospital, especially if it's been more than two days since their symptoms started, it is not so sure if antiviral drugs still help. Clinical research involving patients hospitalized for disease complications is few and of lesser quality. While some indicate that early treatment might be beneficial, there is no scientific agreement about treatment benefits. Therefore, recommendations and antiviral prescription varies between hospitals and physicians.

In Switzerland two antiviral drugs are authorized to treat the flu: Tamiflu® and Xofluza®.

Study aims and methods: The goal of this industry-independent trial is to measure the benefits of Xofluza® compared to placebo (mock medication) in adult patients hospitalized for the flu.

Choice of the medication: The investigators chose Xofluza® instead of Tamiflu® because it is very simple to use (only a single pill instead of twice a day Tamiflu® for 5 days), it has fewer side effects and can be safely given to patients with a wide range of chronic diseases.

Importance: This study is very important because it could lead to a Swiss and international consensus about the utility of antiviral treatment in hospitalized patients.

If beneficial, Xofluza® might be the drug of choice in a future pandemic, when access to a simple to administer and easily stored drug effective at all stages of the illness with few side effects would be of utmost importance.

However, if the trial doesn't show any benefit of Xofluza® administration, antiviral treatment prescription won't be recommended, preserving patients from unneeded medication and from its potential side effects and saving ressources.

Tailoring antiviral use will also help prevent the risk of the virus becoming resistant which might happen in case of overuse.

Patient and public involvement: During the preparation of the study, patient representatives were involved in the development of the research idea, in the discussion concerning its ethical aspects, the feasibility of recruitment, and the selection of questionnaires to measure treatment benefits. They participated in the revision of the lay summary as well. The informed consent form has been developped together with them, in our communication efforts targeting potential participants at the start as well as in the dissemination of the results at the end of the study. Patients representatives also developped together with the investigators the strategy of participants recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participant or participant representative capable of giving signed informed consent.
* Positive reverse transcriptase-polymerase chain reaction (RT-PCR) for influenza A and/or B confirmed on arespiratory tract sample.
* Patient requiring hospitalization.
* National Early Warning Score 2 (NEWS2) of ≥4 at planned randomization

Exclusion Criteria:

* Ongoing pregnancy or breastfeeding (self-reported by the participant or diagnosed by the treating phyisician)
* Known contraindication to baloxavir or to the placebo
* Participant weighing < 40 kg
* Patients already on NAI therapy for the current influenza episode for > 24 hours at the time of randomization.
* Prior treatment with baloxavir for the current influenza epidose
* Immunosuppression defined as 1) cancer treatment with significant negative effect on the immune system; 2) immunosuppressive therapy (treatments comprising a dose of ≥20 mg/day prednisone or equivalent when administered for ≥ 2 weeks, biological therapies, steroid sparing drugs); 3) HIV infection if CD4+ T cell count < 500/µL; 4) organ or stem cell transplantation; 5) patients on the waiting list for a transplant
* Severe underlying respiratory comorbidity requiring long-term oxygenotherapy at home.
* Severe disease requiring ICU care directly at hospitalization.
* Severe hepatic insufficiency or any other severe medical condition when participation in the study puts the patient at risk according to the investigator's judgment.
* History of inclusion in this study during a previous influenza season
* Inclusion in another interventional study with an investigational drug 30 days before inclusion in the study.
* Unability to consent or patient representative unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement | From treatment administration to hospital discharge or NEWS2 score of 2 or lower maintained for 24 h, whichever comes first, assessed up to day 90
  The primary outcome is the time to clinical improvement, calculated from treatment administration, assessed by time to hospital discharge alive or time to a NEWS2 score of 2 or lower maintained for 24 h, whichever comes first.

SECONDARY OUTCOMES:
Clinical status severity score | At 7 days post treatment administration
  A patient's clinical improvement can be assessed by an additional scoring system. Here, a 6-point ordinal scale will be used to capture the different clinical trajectories of the patients (1: discharged; 2: subacute care; 3: acute care without respiratory failure; 4: acute care with respiratory failure; 5: intensive care unit; 6: death) and to measure antiviral treatment's potential benefits with a different tool.
Duration of hospitalization | From treatment administration to hospital discharge, assessed up to day 90
  Duration of hospitalization post-treatment administration, measured in hours
Duration of Oxigen supplementation | From treatment administration to waining of oxygen therapy, assessed up to day 90 (in patients requiring oxygen).
  Duration of O2 supplementation post-treatment administration (in hours).
In-hospital clinical failure | From treatment administration to the end of hospital stay, maximum 30 days after treatment administration
  In-hospital clinical failure, defined as death or ICU or ICMU admission during hospitalization or up to 30 days post treatment administration in case of prolonged hospital stay.
Mortality | From treatment administration during 90 days
  Mortality due to any cause.
Influenza-related complications | From treatment administration during 90 days
  Influenza-related complications, diagnosed by the treating physician (composite outcome defined as pneumonia, sepsis, acute lung injury or ARDS, encephalitis/encephalopathy, myo or -pericarditis, otitis, sinusitis as well as any cardiovascular event (cardiac decompensation, myocardial infarction or stroke))
Antibiotic consumption | From treatment administration to the end of hospital stay, maximum 30 days after treatment administration
  Number of antibiotic days (AD).
Quality of life | At day 90-days post treatment administration
  Impact of antiviral treatment on patient quality of life after discharge using the EQ-5D-5L scale (5-level EQ-5D version).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Viral shedding | On day 3 after treatment administration.
  Number of participants with detectable RNA in respiratory sample on day 3 after treatment administration.
Duration of infectious viral shedding | On day 3 post-treatment administration
  Infectious viral load in respiratory sample at day 3 post-treatment administration.

OTHER OUTCOMES:
Serious adverse events, SAR and SUSAR | From treatment administration to the end of hospital stay, maximum 30 days after treatment administration
  Safety outcomes will be SAE unrelated to the natural history of influenza, SAR and SUSAR.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Vetter, MD, Principal Investigator — University Hospital, Geneva; Nicolas Muller, Professor, Principal Investigator — Department of Infectious Diseases and Hospital epidemiology, University Hospital Zürich; Matteo Mombelli, MD, Principal Investigator — Department of internal medicine, Locarno Regional Hospital EOC; Oriol Manuel, Pr, Principal Investigator — Center for organ transplantation, Lausanne University Hospitals
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). IPD can be shared with investigators whose proposed use of the data has been approved by an independent review committee, for, as an example, individual participant data meta-analysis. The approval of the biobank regulation committee, which includes the coordinating PI, the sites PI and the responsibles of the biobank is also required on a case by case basis.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and up to 10 years after publication.
Access Criteria: IPD can be shared with investigators whose proposed use of the data has been approved by an independent review committee. The approval of the biobank regulation committee, which includes the coordinating PI, the sites PI and the responsibles of the biobank is also required on a case by case basis.

REFERENCES:
- [Background] Hosszu-Fellous K, Vetter P, Agoritsas T, Kaiser L. Which trial do we need? Randomized, placebo-controlled trial of antiviral treatment in patients hospitalized for influenza. Clin Microbiol Infect. 2024 May;30(5):567-569. doi: 10.1016/j.cmi.2024.01.025. Epub 2024 Feb 3. No abstract available. PMID 38316358
- [Derived] Hosszu-Fellous K, Poncet A, Cabecinhas ARG, Schibler M, Meyer B, Prendki V, Huttner A, Carballo S, Pouillon M, Slankamenac K, Bart PA, Bernasconi E, Manuel O, Mombelli M, Mueller NJ, Kaiser L, Vetter P. Antiviral treatment in adult patients hospitalized for influenza: study protocol for a multi-center, randomized, placebo-controlled trial on the efficacy of baloxavir marboxil to reduce time to clinical improvement and the risk for severe complications (the INFLUENT trial). Trials. 2025 Nov 24;26(1):538. doi: 10.1186/s13063-025-09248-0. PMID 41286959